CLINICAL TRIAL: NCT04025489
Title: Randomized Control Trial of Vitamin D Supplementation on Surrogate Markers of Ageing, Association/Interactions With Selected Ageing-related Genes, Glycemic and Metabolic Markers in North Indian Individuals With the Prediabetes
Brief Title: Vitamin D Supplementation on Surrogate Markers of Ageing, Ageing Genes, Glycemic and Metabolic Markers in North India
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diabetes Foundation, India (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Presidant, Diabetes Foundation, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DFI
Record Dates: First submitted 2019-05-15; First posted 2019-07-19 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-07

CONDITIONS: Vitamin D Supplementation; PreDiabetes; Aging
Keywords: Pre-diabetes; Type 2 Diabetes; Genes; Supplementation
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D and Placebo (Experimental): Doses of cholecalciferol (commercial name, Calcirol) 60,000IU (sachets, dissolved in half glass milk) once per week for eight weeks to intervention group and placebo (Lactose Granules) to the placebo group according to the random numbers generated by the computer.
  Interventions: Dietary Supplement: Randomized control trial of vitamin D supplementation

INTERVENTIONS:
Dietary Supplement: Randomized control trial of vitamin D supplementation — This open-label randomized placebo-controlled prospective trial will be randomized into two groups; lifestyle modification counseling along with intervention with either vitamin D or placebo. Anthropometry, body composition, levels of vitamin D, blood glucose (including oral glucose tolerance test) and dietary assessments will be assessed periodically (every 3 months). In those having recurrent vitamin D deficiency, the course of vitamin D will be repeated. Diet and exercise will be recommended as per the regular norms for overweight and obese subjects. Clinical and dietary profile, sunlight exposure, glycemic and lipid profile other metabolic parameters, body composition, hand grip strength, leukocyte telomerase length and telomerase activity will be assessed at enrolment time and one-year intervention. As mentioned above, genes related to ageing will be evaluated. Effects on polymorphisms of pro-ageing genes will be assessed.

SUMMARY:
Prediabetes is a substantial problem in India not only because it itself can be associated with morbidities such as coronary artery disease but also because it is a point of important for prevention of diabetes. It is not clear if apparent accelerated aging in Indian population associated with heightened tendency for prediabetes, metabolic syndrome, atherosclerosis and dys-metabolic state etc. could, besides lifestyle factors, be related to vitamin D deficiency, or ageing-related genes, or interaction between the two. This study is based on the assumption that the supplementation of vitamin d could lead to reversal to normal glucose regulation and may slow aging process in individuals with pre-diabetes.

DETAILED DESCRIPTION:
Asian Indians develop metabolic syndrome and diabetes earlier than in most population. In other words, Asian Indians have all the risk factors which may predispose to accelerated ageing; insulin resistance, dysglycemia, subclinical inflammation, and vasculopathy.

Vitamin D deficiency is widespread in both urban and rural populations of India. It is possible that vitamin D may also act on pathway related to aging which also are common to chronic diseases like diabetes. In this respect the surrogate markers of ageing (leukocyte telomerase length and telomerase activity) could be affected if vitamin D deficiency occurs. While some studies have shown relationship between vitamin D supplementation and leukocyte telomerase length in other populations, such study has not been systematically performed in Asian Indians. In this context, it is also not clear if some proposed genes of ageing may have some influence of development of prediabetes or diabetes and may interact with vitamin D. One of the candidate gene MSTN, according to our previous study, showed close correlation with excess body fat and decrease muscle mass, body composition characteristics conducive to development of diabetes. Additionally, deficiency of vitamin D could be linked to insulin resistance, prediabetes, though these issues have been debated. Some studies suggest that vitamin D supplementation may improve insulin sensitivity in Asian Indians. A research focusing on relationship of vitamin D supplementation with pro-ageing metabolic factors (glycemia, insulin resistance etc,), ageing related genes and surrogate markers of ageing is needed.

This study has two components; cross-sectional and prospective. Cross-sectional study will be of 2 years duration where 500 subjects from urban area of Delhi will be screened randomly for the vitamin D deficiency and its determinants including duration of sun exposure. The population will be representative of different socio-economic strata of the society. In this, vitamin D levels, leukocyte telomerase length and telomerase activity in peripheral blood leukocytes, telomerase activity and single nucleotide polymorphisms [ACTN3, VDR, FOXO3A, SIRT1 and MSTN] in prediabetes Asian Indians.

Second part consists of open-label randomized placebo-controlled prospective trial, in which the investigators would be enrolling 200 prediabetic subjects with vitamin D deficiency. These subjects will be randomized into two groups; lifestyle modification counseling along with intervention with either vitamin D or placebo. Anthropometry, body composition, levels of vitamin D, blood glucose (including oral glucose tolerance test) and dietary assessments will be assessed periodically (every 3 months). In those having recurrent vitamin D deficiency, the course of vitamin D will be repeated. Diet and exercise will be recommended as per the regular norms for overweight and obese subjects. Clinical and dietary profile, sunlight exposure, glycemic and lipid profile other metabolic parameters, body composition, hand grip strength, leukocyte telomerase length and telomerase activity will be assessed at enrolment time and one year intervention. As mentioned above, genes related to ageing will be evaluated. Appropriate statistical methods will be used to see effects of intervention with Vitamin D on metabolic state (particularly insulin resistance and glycemia) and leukocyte telomerase length and telomerase activity. Effects of polymorphisms of pro-ageing genes will be assessed

ELIGIBILITY:
Inclusion and Exclusion Criteria of Cross Sectional and Prospective Study:

Cross-sectional Study:

Inclusion Criteria: Individuals with prediabetes, aged 20-60 years.

Exclusion Criteria:

1. Received Vitamin D or calcium supplementation in the previous six months.
2. On any medication within last one month which could potentially influence insulin secretion, insulin sensitivity, vitamin D or calcium metabolism and on any medication that activate steroid and xenobiotic receptors, and drugs used in transplantation.
3. Severe end organ damage or chronic diseases: renal/hepatic failure, any malignancy, major systemic illness etc.
4. Known case of diabetes mellitus, HIV infection and other endocrine disorders.

Prospective Intervention Study:

Design: Randomized open labeled placebo-controlled trial.

Inclusion Criteria:

1. Pre-diabetes:

   1. Fasting blood glucose ≥100mg/dl and <125.99mg/dl, or
   2. 2-h plasma glucose ≥140mg/dl and <200mg/dl (after ingestion of 75 g anhydrous oral glucose), and
2. Baseline blood level of 25 hydroxy vitamin D <30ng/dl.
3. Aged 20-60 years

Exclusion Criteria:

1. Received Vitamin D and/or calcium supplementation in the previous six months.
2. On any medication within last one month which could potentially influence insulin secretion, insulin sensitivity, vitamin D or calcium metabolism (e.g. metformin, thiazolidinediones, steroids etc) and on any medication that activate steroid and xenobiotic receptor and drugs used in transplantation (e.g. steroids, calcitonin etc.)
3. Severe end organ damage or chronic diseases: renal/ hepatic failure, any malignancy, nephrotic syndrome, malabsorption etc.
4. Known case of HIV infection.
5. Primary or tertiary hyperparathyroidism, granulomatous disorders (e.g. sarcoidosis) and any lymphomas.
6. Known case of diabetes mellitus.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Investigation of gene polymorphism and other markers in 500 subjects | 1 year
  single nucleotide polymorphisms [ACTN3, VDR, FOXO3A, SIRT1 and MSTN] Asian Indians with prediabetes.

SECONDARY OUTCOMES:
Effect of vitamin d supplementation on raging and other metabolic measures. | 2 year
  Vitamin D supplementation could Improve insulin action and glucose physiology, leading to lowering of blood glucose levels in persons with prediabetes.
  1. Increase/preserve leucocyte telomerase length and activity, thus having positive effects on ageing.
  2. Improve insulin action and glucose physiology, leading to lowering of blood glucose levels in persons with prediabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- Fortis-C-DOC Centre of Excellence for Diabetes, Metabolic Diseases and Endocrinology, Delhi, India

IPD SHARING:
Plan to Share IPD: No
This study will be conducted at the outpatient department of National Diabetes, Obesity and Cholesterol Foundation (N-DOC), Diabetes Foundation (India) (DFI) and Fortis-C-DOC, Centre of Excellence for Diabetes, Metabolic Diseases and Endocrinology, New Delhi, India.